CLINICAL TRIAL: NCT01962155
Title: Prospective Stuy in Evaluating Hepatic Fibrosis Related to Hepatitis B Virus
Brief Title: Prospective Stuy in Evaluating Hepatic Fibrosis Related to Hepatitis B Virus Using Non-invasive Parameters
Acronym: HBV
Status: Completed | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Guiqiang Wang, MD, Peking University First Hospital
Other Study IDs: 2013ZX10002005
Record Dates: First submitted 2013-10-05; First posted 2013-10-14 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Hepatitis B; Liver Fibrosis
Keywords: Fibrosis; Liver Cirrhosis; non-invasive; biopsy; hepatitis B virus
MeSH Terms: conditions — Hepatitis B; Liver Cirrhosis; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — liver biopsy samples and blood samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- chronic infected with hepatitis B virus: patients infected with hepatitis B virus for at least 6 months and agreed with liver biopsy

SUMMARY:
The aim of our prospective study is to construct and validate a non-invasive model consisting biochemical markers, FibroScan, and radiological parameters for evaluating liver fibrosis caused by hepatitis B virus in mainland China.

DETAILED DESCRIPTION:
Up to Oct, 2015,total of 1800 patients with chronic HBV infection were enrolled. Paired blood and liver biopsy samples were collected. Blood samples stored at -80 degree Celsius. Liver biopsy samples were judged by three pathology experts.

ELIGIBILITY:
Inclusion Criteria:

1. HBsAg positive for at least 6 months
2. agree to have liver biopsy
3. Male or female aged 18 to 65 years old

Exclusion Criteria:

1. Patients with alcoholic liver disease, autoimmune liver disease, heretic liver disease, drug induced liver disease,nonalcoholic liver disease or other chronic liver disease
2. platelet count < 80000/L
3. prothrombin activity ≤ 60%
4. patients with any disease or condition which the investigator or treating physician feels would interfere with the trial or the safety of the subject

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients infected with hepatitis B virus for at least 6 months
Sampling Method: Probability Sample
Enrollment: 1841 (Actual)
Dates: Start 2013-08; Primary Completion 2015-12 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
determine whether a non-invasive test or a combination of non invasive tests may be used to accurately evaluate liver fibrosis in patients with chronic hepatitis B | singular evaluation at the time of liver biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Guiqiang Wang, Principal Investigator — Peking University First Hospital
Locations (30):
- China (30):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - 302 Military Hospital of China, Beijing, Beijing Municipality
  - Beijing Ditan Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Southwest Hospital, Third Military Medical University, Chongqing, Chongqing Municipality
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Guangzhou Eighth People's Hospital, Guangzhou, Guangdong
  - The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - The Third people's Hospital of Shenzhen, Shenzhen, Guangdong
  - The People's Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - The Third People's Hospital of Qinhuangdao, Qinhuangdao, Hebei
  - The Third Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South Hospital, Changsha, Hunan
  - 81 Military Hospital of China, Nanjing, Jiangsu
  - The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu
  - The Second Hospital of Nanjing, Nanjing, Jiangsu
  - Dalian the Sixth People's Hospital, Dalian, Liaoning
  - The Sixth People's Hospital of Shenyang, Shenyang, Liaoning
  - Yantai City Hospital for Infectious Diseases, Yantai, Shandong
  - Shan Xi Medical University, Taiyuan, Shanxi
  - Zhejiang First Hospital, Hangzhou, Zhejiang
  - Beijing Youan Hospital, Capital Medical University, Beijing
  - China-Japan Friendship Hospital, Beijing
  - The 305 Hospital of People's Liberation Army, Beijing
  - West China Hospital, Sichuan University, Chengdu
  - Shanghai Public Health Clinical Center, Shanghai
  - Shanghai Ruijin Hospital, Shanghai

REFERENCES:
- [Derived] Li J, Dong XQ, Cao LH, Zhang ZQ, Zhao WF, Shang QH, Zhang DZ, Ma AL, Xie Q, Gui HL, Zhang G, Liu YX, Shang J, Xie SB, Liu YQ, Zhang C, Wang GQ, Zhao H; China HepB Related Fibrosis Assessment Research Group. Factors associated with persistent positive in HBV DNA level in patients with chronic Hepatitis B receiving entecavir treatment. Front Cell Infect Microbiol. 2023 Jun 16;13:1151899. doi: 10.3389/fcimb.2023.1151899. eCollection 2023. PMID 37396307
- [Derived] Li J, Wu Z, Wang GQ, Zhao H. Hepatitis B core-related antigen reflects viral replication and protein production in chronic hepatitis B patients. Chin Med J (Engl). 2021 Mar 17;134(10):1160-1167. doi: 10.1097/CM9.0000000000001418. PMID 33734135
- [Derived] Li J, Dong XQ, Wu Z, Ma AL, Xie SB, Zhang XQ, Zhang ZQ, Zhang DZ, Zhao WF, Zhang G, Cheng J, Xie Q, Li J, Zou ZQ, Liu YX, Wang GQ, Zhao H; China Hepatitis B Related Fibrosis Assessment Research Group. Unsatisfying antiviral therapeutic effect in patients with mother-to-child transmissed chronic hepatitis B virus infection: a prospective multi-center clinical study. Chin Med J (Engl). 2019 Nov 20;132(22):2647-2656. doi: 10.1097/CM9.0000000000000522. PMID 31725459
- [Derived] Deng Y, Zhao H, Zhou J, Yan L, Wang G; China HepB-Related Fibrosis Assessment Research Group. Angiopoietin-like protein as a novel marker for liver fibrosis in chronic hepatitis B patients with normal to minimally raised ALT. BMC Infect Dis. 2017 Sep 29;17(1):650. doi: 10.1186/s12879-017-2728-7. PMID 28962551